CLINICAL TRIAL: NCT07405164
Title: A Multicenter, Open-label, Phase 3 Extension Study to Evaluate the Long-term Efficacy and Safety in Participants Who Are Currently on Treatment in a Belzutifan Study (LITESPARK-043)
Brief Title: Extension Study for Participants in Studies That Include Belzutifan (MK-6482-043/LITESPARK-043)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-043; U1111-1325-4582 (Registry Identifier: UTN); 2025-524160-38-00 (Registry Identifier: EU CT); MK-6482-043 (Other: MSD)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Von Hippel-Lindau Disease; Carcinoma, Renal Cell
MeSH Terms: conditions — von Hippel-Lindau Disease; Carcinoma, Renal Cell | interventions — belzutifan; palbociclib; Nivolumab; lenvatinib; cabozantinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Belzutifan Monotherapy (Experimental): Participants on active treatment assigned to belzutifan monotherapy in a parent study are transitioned to this extension study. Participants will continue the same dose and frequency of intervention as they were receiving in the parent study at the time of the transition. Treatment will continue until progressive disease (PD), unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Interventions: Drug: Belzutifan
- Cohort B: Belzutifan Combination Therapy (Experimental): Participants on active treatment assigned to a belzutifan combination therapy in a parent study are transitioned to this extension study. Participants will continue the same dose and frequency of intervention as they were receiving in the parent study at the time of the transition. Treatment will continue until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Interventions: Drug: Belzutifan; Drug: Palbociclib; Drug: Nivolumab; Drug: Lenvatinib; Drug: Cabozantinib
- Cohort C: Non-Belzutifan Therapy (Active Comparator): Participants on active treatment assigned to a non-belzutifan therapy in a parent study are transitioned to this extension study. Participants will continue the same dose and frequency of intervention as they were receiving in the parent study at the time of the transition. Treatment will continue until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Interventions: Drug: Lenvatinib; Drug: Cabozantinib; Drug: Everolimus

INTERVENTIONS:
Drug: Belzutifan — Belzutifan is administered orally at 120 mg once daily (qd) OR 160 mg twice daily (bid) OR 160 mg three times daily (tid) OR 200 mg qd OR 240 mg qd until progressive disease (PD), unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Other Names: MK-6482, PT2977, WELIREG
  Arms: Cohort A: Belzutifan Monotherapy; Cohort B: Belzutifan Combination Therapy
Drug: Palbociclib — Palbociclib is administered orally at 75 mg qd OR 100 mg qd OR 125 mg qd for 21 consecutive days; 7 days off, until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Arms: Cohort B: Belzutifan Combination Therapy
Drug: Nivolumab — Nivolumab is administered intravenously at 480 mg until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Arms: Cohort B: Belzutifan Combination Therapy
Drug: Lenvatinib — Lenvatinib is administered orally at 20 mg qd until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Arms: Cohort B: Belzutifan Combination Therapy; Cohort C: Non-Belzutifan Therapy
Drug: Cabozantinib — Cabozantinib is administered orally at 60 mg qd until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Arms: Cohort B: Belzutifan Combination Therapy; Cohort C: Non-Belzutifan Therapy
Drug: Everolimus — Everolimus is administered orally at 10 mg qd until PD, unacceptable toxicity, withdrawal of consent, death, investigator decision, or study termination.
  Arms: Cohort C: Non-Belzutifan Therapy

SUMMARY:
Researchers are looking for new ways to treat advanced solid tumors and von Hippel-Lindau (VHL)-related tumors:

* Advanced means the cancer has spread to other parts of the body (metastatic) or cannot be removed with surgery
* Solid tumors are cancers mostly in body organs and tissues, not in the blood or other body liquids
* VHL-related tumors are tumors caused by VHL disease. VHL disease is passed down from parents to children and people with VHL disease have a higher chance of getting certain types of cancer

Researchers want to learn about the long-term effects of a trial medicine called belzutifan. Belzutifan, also called MK-6482, is designed to block a protein that helps tumors grow and survive. This is an extension trial, which means only people who were in certain other belzutifan trials (called parent trials) may be able to join. The goal of this trial is to learn how long people live after they start taking belzutifan.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Participants with advanced solid tumors or von Hippel-Lindau-related neoplasms who are participating in belzutifan-containing studies and on active treatment in a belzutifan parent study.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has an on-going serious adverse event in the parent study, unless no longer hospitalized and considered clinically stable.
* Is currently on a dose interruption due to an Adverse Event (AE) in the parent study; once treatment has been resumed in the parent study, the participant is eligible to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-03-11 (Estimated); Primary Completion 2034-01-14 (Estimated); Study Completion 2034-01-14 (Estimated)

PRIMARY OUTCOMES:
Cohort A and Cohort B: Overall Survival (OS) | Up to approximately 7 years
  Overall survival is defined as the time from randomization or the first dose of any study intervention in the parent study to death due to any cause.

SECONDARY OUTCOMES:
Number of Participants Who Experience One or More Adverse Events (AE) | Up to approximately 2 years
  An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Number of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 2 years
  An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/